CLINICAL TRIAL: NCT06754319
Title: Pathogenesis of Pediatric Obsessive-compulsive Disorder: Based on the Microbiota-gut-brain Axis
Status: Enrolling by invitation | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Other Study IDs: SMHC-POCD-001
Record Dates: First submitted 2024-12-15; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-11

CONDITIONS: Obsessive-Compulsive Disorder; Tic Disorder
Keywords: microbiota-gut-brain axis; pediatric OCD; microbiome
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Tic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fecal, blood, brain MRI and EEG
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- pediatric OCD patients: Drug-naïve or drug-free pediatric patients with OCD will be enrolled in this group. After data collection, they will receive treatment with SSRIs.
- pediatric OCD patients comorbid with TD: Drug-naïve or drug-free pediatric OCD patients comorbid with TD will be enrolled in this group. After data collection, they will receive treatment with SSRIs and antipsychotics.
- healthy controls: Healthy children and adolescents will be enrolled in this group for data collection.

SUMMARY:
This study aims to investigate the characteristics of the microbiota-gut-brain axis in pediatric patients with obsessive-compulsive disorder (OCD) through performing an integrated analysis of gut microbiota, serum metabolomics, neuroimaging and electroencephalography (EEG), conducted before and after treatment with selective serotonin reuptake inhibitors (SSRIs). The results will be compared with those of pediatric OCD paitents comorbid with tic disorder (TD) and healthy controls. The findings are expected to further elucidate the potential pathogenesis of OCD, providing a theoretical basis for identifying novel clinical intervention targets and optimizing treatment strategies.

ELIGIBILITY:
We recruited outpatient children and adolescents with OCD confirmed by the Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (4th edition). The following inclusion and exclusion criteria were also applied:

Inclusion Criteria:

(1) 7-17 years old, (2) Y-BOCS score ≥16, (3) with or without a history of TD, (4) Drug-naïve or drug-free for 8 weeks, (5) Wechsler IQ score ≥ 80.

Exclusion Criteria:

* History of serious medical, neurological illness or other psychotic disorders other than OCD (tic disorder excepted).
* Previous exposure to cognitive behavioral therapy (CBT) for OCD or TD.
* serious suicide risk.
* Has taken antibiotics, probiotics, prebiotics, corticosteroids, nonsteroidal anti-inflammatory drugs (NSAIDs), or immunosuppressants within the past 8 weeks.
* Has a history of gastrointestinal diseases such as inflammatory bowel disease, irritable bowel syndrome, constipation, hemorrhoids, or a history of gastrointestinal surgery, or has a history of autoimmune diseases such as rheumatoid arthritis or systemic lupus erythematosus.
* Participants with claustrophobic, heart pacemaker, mechanical heart valve, mechanical implant such as an aneurysm clip, hip replacement, or any other pieces of metal that have accidentally entered their body.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Drug-naïve or drug-free pediatric patients with OCD, drug-naïve or drug-free pediatric OCD patients comorbid with TD, and healthy control.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-08-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the diversity and composition of the microbiome before and after drug treatment. | Before and after treatment with SSRIs for 12 weeks
  The diversity (including alpha-diversity and beta-diversity) and composition will be measured in OCD patients and OCD patients with TD before and after drug treatment, and the results will be compared with those of healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD, MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China